CLINICAL TRIAL: NCT06043349
Title: Effectiveness and Safety of Platelet-rich Plasma and Topical 5% Minoxidil Combination Compared to Topical 5% Minoxidil Monotherapy in Male Androgenetic Alopecia
Brief Title: Effectiveness and Safety of Platelet-rich Plasma and Topical 5% Minoxidil Combination in Male Androgenetic Alopecia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Adhika Ayu Lestari, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23020292
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Androgenetic Alopecia
Keywords: Platelet-Rich Plasma; Topical Minoxidil; Combination Therapy
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Intervention Model Description: This study is a controlled clinical trial on male androgenetic alopecia. Research subjects will be randomly divided into two groups. The first group will receive a combination therapy of PRP injection and topical 5% minoxidil, while the second group will receive topical 5% minoxidil as monotherapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The first group, called the intervention group, will receive a combination therapy of platelet-rich plasma injection (PRP) with topical 5% minoxidil for three months. PRP injection will be given every 4 weeks with a total of three injections. Respondents will be instructed to apply topical minoxidil twice daily for three months.
  Interventions: Combination Product: Platelet-Rich Plasma and Topical 5% Minoxidil
- Control Group (Active Comparator): The second group (control group) will receive topical 5% minoxidil as standard therapy. Respondents will be instructed to apply topical minoxidil twice daily for three months.
  Interventions: Drug: Topical 5% Minoxidil

INTERVENTIONS:
Combination Product: Platelet-Rich Plasma and Topical 5% Minoxidil — The intervention group will receive three PRP injections during three months in addition to the topical 5% minoxidil.
  Arms: Intervention Group
Drug: Topical 5% Minoxidil — The intervention group will receive topical 5% minoxidil as standard therapy for male androgenetic alopecia.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn about the effectiveness and safety of platelet-rich plasma (PRP) and topical 5% minoxidil combination therapy compared with topical 5% minoxidil monotherapy in male androgenetic alopecia.

The main questions it aims to answer are:

* Is there a difference in average change of hair density between groups that were given a combination of PRP injection and topical minoxidil compared to topical minoxidil as monotherapy?
* Is there a difference in average change of hair thickness between groups that were given a combination of PRP and topical minoxidil compared to topical minoxidil as monotherapy?
* Are there any differences in side effects between groups that were given combination of PRP and topical minoxidil compared to topical minoxidil as monotherapy?

DETAILED DESCRIPTION:
The trial will be held for three months in Jakarta, Indonesia. Participants are required to undergo hair examinations every 4 weeks, for a total of 4 visits. Researchers will compare groups that were given a combination of PRP and topical minoxidil compared to topical minoxidil alone as a control group. Hair density, hair thickness, and overall side effects of treatment will be measured at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 50 years old
* Diagnosed with grade III-VI androgenetic alopecia based on Hamilton-Norwood scale
* Willing to be the research subject and make regular follow-up visits.

Exclusion Criteria:

* Conditions of baldness other than androgenetic alopecia based on anamnesis and physical examination, namely telogen effluvium, alopecia areata, trichotillomania, syphilis secondary, systemic lupus erythematosus, alopecia due to chemotherapy, autoimmune, or malignancy.
* Taking oral medications or vitamins that aim to increase the amount of hair in the last 1 month.
* Using topical medication that aims to increase the amount of hair in the last 2 weeks.
* Suffering from active bacterial, viral, or fungal infections of the scalp.
* Underwent cosmetic procedures for androgenetic alopecia treatment (such as PRP injections, laser procedures, or microneedle) within the last 3 months prior to the study.
* History of keloids.
* History of blood clotting disorders.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male patient with androgenetic alopecia
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Hair Density | Three months
  Change in average hair density will be reported in /cm2
Hair Thickness | Three months
  Change in average hair thickness will be reported in milimeters

SECONDARY OUTCOMES:
Subjective side effects | Three months
  The patients subjective side effects from both intervention and control group will be reported using questionnaire during follow-up visits. Subjective side effects which will be reported consist of pain, itch, and burning sensation. Each subjective complaint will be reported as "Yes" or "No". Other subjective side effects, if any, will also be noted under the term "Other".
Objective side effects | Three months
  Researcher will report any objective side effects found during follow-up visits. The main objective side effects that will be reported are erythema and hypertrichosis. Each finding will be reported as "Yes" or "No". Other objective side effects, if any, will be noted under the term "Other".

CONTACTS AND LOCATIONS:
Overall Officials: Adhika A Lestari, MD, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (1):
- Dr. Cipto Mangunkusumo National General Hospital, Jakarta Pusat, Greater Jakarta Area, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elena EP, Irina OS. Combination therapy with platelet-rich plasma and minoxidil leads to better clinical results than monotherapy with these methods in men with androgenetic alopecia. Int J Trichology. 2022 Jan-Feb;14(1):1-7. doi: 10.4103/ijt.ijt_50_19. Epub 2022 Feb 1. PMID 35300100
- [Result] Singh SK, Kumar V, Rai T. Comparison of efficacy of platelet-rich plasma therapy with or without topical 5% minoxidil in male-type baldness: A randomized, double-blind placebo control trial. Indian J Dermatol Venereol Leprol. 2020 Mar-Apr;86(2):150-157. doi: 10.4103/ijdvl.IJDVL_589_18. PMID 31823902